CLINICAL TRIAL: NCT01680055
Title: Collection of Blood and Bone Marrow From Patients With Aplastic Anemia for Analysis of Adhesion Molecules, Chemokines and Their Receptors
Status: Withdrawn | Type: Observational
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Director, Shandong University
Other Study IDs: Aplastic Anemia 1
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2012-09

CONDITIONS: Aplastic Anemia; Healthy
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- AA-ATG: Acquired Aplastic Anemia Patients Treated with Antithymocyte Globulin plus Cyclosporine

SUMMARY:
This study is designed to collect bone marrow and/or peripheral blood cells and plasma, for the analysis of adhesion molecules, chemokines and their receptors from newly-diagnosed aplastic anemia patients, and patients treated with antithymocyte globulin plus cyclosporine

ELIGIBILITY:
Inclusion Criteria:

* patients who fulfilled entry criteria of acquired aplastic anemia age range 16-70 years

Exclusion Criteria:

* Patients complicated with diabetes, tumor, pregnancy, active infection, or connective tissue diseases, such as systemic lupus erythematosus.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Aplastic Anemia
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02; Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
hematologic response | 6 months following antithymocyte globulin plus cyclosporine treatment
  hematologic response at 6 months following antithymocyte globulin plus cyclosporine treatment, defined as no longer meeting the criteria for severe aplastic anemia

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China